CLINICAL TRIAL: NCT02729038
Title: A Phase I, Open-Label, Single-Dose, Multi-Part Study to Assess the Pharmacokinetics of Gepotidacin (GSK2140944) in Male and Female Adult Subjects With Varying Degrees of Renal Impairment and in Matched Control Subjects With Normal Renal Function
Brief Title: Pharmacokinetic Study of Gepotidacin in Subjects With Varying Degrees of Renal Impairment and in Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116849
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Infections, Bacterial
Keywords: Normal Renal Function; end stage renal disease (ESRD); Pharmacokinetics; Gepotidacin; Renal Impairment
MeSH Terms: conditions — Bacterial Infections; Kidney Failure, Chronic; Renal Insufficiency | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1: Subjects with normal renal function (Group A) (Experimental): Subjects with normal renal function will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion.
  Interventions: Drug: Gepotidacin
- Part 1: subjects with moderate renal impairment (Group B) (Experimental): Subjects with moderate renal impairment will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion.
  Interventions: Drug: Gepotidacin
- Part 1: subjects with severe renal impairment (Group C) (Experimental): Subjects with severe renal impairment and subjects with ESRD not on hemodialysis will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion.
  Interventions: Drug: Gepotidacin
- Part 2: subjects with normal renal function (Group D) (Experimental): Subjects with normal renal function will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion.
  Interventions: Drug: Gepotidacin
- Part 2: subjects with mild renal impairment (Group E) (Experimental): Subjects with mild renal impairment will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion.
  Interventions: Drug: Gepotidacin
- Part 2: subjects with ESRD on hemodialysis (Group F) (Experimental): Subjects with ESRD on hemodialysis will receive a single dose of gepotidacin 750 mg administered as a 2 hour IV infusion starting approximately 2 hours before the initiation of the last hemodialysis session of the week (Period 1) and gepotidacin 750 mg administered as a 2 hour IV infusion starting within 2 hours after completion of the last hemodialysis session of the week (Period 2).
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin after reconstitution is a clear, dark brown to dark brownish-yellow solution, free from visible particulate matter. Subjects will receive gepotidacin 750 mg single IV dose over 2 hours.

SUMMARY:
This study will be conducted to determine if altered renal function affects the plasma pharmacokinetics of gepotidacin, which will inform if dosing recommendations based upon renal impairment are required. The objective of this study is to compare the pharmacokinetics of gepotidacin administered as a 750 milligram (mg) intravenous (IV) dose in normal healthy subjects compared with subjects with mild, moderate, and severe renal impairment, and with subjects with end stage renal disease (ESRD). This is a Phase I, nonrandomized, open-label, parallel-group, multi-center, multi-part study. In Part 1, up to 16 subjects with normal renal function will be matched to approximately 8 subjects with moderate renal impairment, and approximately 8 subjects with severe renal impairment and/or subjects with ESRD not on hemodialysis for a total of approximately 32 subjects. In Part 2 (optional), approximately 4 to 8 subjects with normal renal function (if enrolled), approximately 4 to 8 subjects with mild renal impairment, and approximately 4 to 8 subjects with ESRD on hemodialysis will be enrolled for a total of approximately 12 to 24 subjects. The duration from Screening to the Follow-up Visit will be approximately 44 days for Part 1 and approximately 50 days for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Age: Male or female subject between 18 and 80 years of age, inclusive.
* Healthy subject must be in clinically stable health as determined by the investigator based on medical history, clinical laboratory results (serum chemistry, hematology, urinalysis, and serology), vital sign measurements, 12 lead ECG results, and physical examination findings. Subject with renal impairment must have clinical laboratory values consistent with their disease and are approved by the investigator.
* Subject with renal impairment (mild, moderate, severe, or subjects with ESRD) may be taking medications, which in the opinion of the investigator, are believed to be therapeutic but do not affect study drug absorption, distribution, metabolism, or excretion. These medications must be stable doses taken for at least 7 days before the first dose of study drug.
* Subject with normal renal function or renal impairment (estimated Glomerular Filtration Rate [eGFR] corresponding to the calculated eGFR [the estimated eGFR may be rounded to the nearest integer]) at Screening.
* Subjects with ESRD on hemodialysis should be on hemodialysis for at least 3 months before Screening and is able to tolerate a hemodialysis treatment lasting 3 to 4 hours with blood flow rates of >200 milliliter (mL)/minute (min).
* Alanine aminotransferase (ALT) and bilirubin <1.5 × upper limit of normal (ULN; isolated bilirubin >1.5 × ULN is acceptable, if bilirubin is fractionated and direct bilirubin <35%).
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18.5 and 40 kg/square meter (m^2), inclusive.
* Male or Female. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies:

Nonreproductive potential defined as:

* Premenopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, or Documented bilateral oophorectomy
* Postmenopausal defined as 12 months of continuous spontaneous amenorrhea (in questionable cases a blood sample will be obtained to test for simultaneous follicle-stimulating hormone) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

Reproductive potential and agrees to follow 1 of the options listed in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential requirements from 30 days prior to the first dose until completion of the Follow-up Visit.

For subjects with indeterminate pregnancy test results or a persistently low human chorionic gonadotropin results, nonpregnancy status must be documented by other means (subjects with ESRD only).

* Capable of giving signed informed consent as described in protocol, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Subject has a clinically significant abnormality in past medical history or at the Screening physical examination (excluding renal insufficiency and other related stable medical conditions within the renally impaired population of subjects [e.g., hypertension, diabetes, or anemia, which should be stable for at least 3 months before the first dose of study drug]) that in the investigator's opinion may place the subject at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current cardiac, hepatic, neurologic, gastrointestinal (GI), respiratory, hematologic, or immunologic disease.

Subject has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the subject at risk, in the opinion of the investigator.

* Subject has a functioning renal transplant.
* Subject with renal impairment has a systolic blood pressure outside the range of 90 to 200 millimeter of mercury (mm Hg), a diastolic blood pressure outside the range of 45 to 110 mm Hg, or a heart rate outside the range of 40 to 120 beats per minute (bpm).
* Subject with renal impairment has a hemoglobin value <9 grams (g)/decilitre (dL).
* Female subject has a positive pregnancy test result or is lactating at Screening or upon admission to the clinic.
* Use of a systemic antibiotic within 30 days of Screening
* Within 2 months before Screening, either a confirmed history of Clostridium difficile diarrhoea infection or a past positive Clostridium difficile toxin test.
* Subject has a history of drug and/or alcohol abuse within 6 months before Screening, as determined by the investigator, or subject has a positive drug screen at Screening or upon admission to the clinic. For subjects with renal impairment, a positive drug screen result related to the use of prescription medications is allowed per investigator review and approval, and tetrahydrocannabinol use is allowed per investigator review and approval.
* History of sensitivity to any of the study drugs, components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) medical monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain IV cannula patency).
* Subject has used medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) or competitors of renal tubular secretion (e.g., probenecid) within 30 days before dosing.
* Subjects cannot use any over-the-counter, or prescription medication (except for hormonal contraceptives and/or acetaminophen), vitamin supplement, or herbal medication within 7 days (or 5 half-lives, whichever is longer) before dosing and during the study within 7 days before dosing and during the study.
* Subjects with normal renal function have a presence of hepatitis B surface antigen or positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study treatment. A subject with renal impairment with stable hepatitis C who has normal liver function test results is allowed with investigator approval.
* A positive test for human immunodeficiency virus antibody.
* Subject has clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at Screening or Day -1 (and Day 7 for Group F only), other than those associated with underlying renal conditions or other stable medical conditions consistent with the disease process.
* Subject with normal renal function has a baseline corrected QT interval using the Fridericia formula (QTcF) of >450 milliseconds (msec) and subject with renal impairment has a baseline QTcF of >480 msec.
* Donation of blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Previous exposure to gepotidacin within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subject is unable to comply with all study procedures, in the opinion of the investigator.
* The subject should not participate in the study, in the opinion of the investigator or Sponsor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20385

REFERENCES:
- [Background] Hossain M, Tiffany C, Raychaudhuri A, Nguyen D, Tai G, Alcorn H Jr, Preston RA, Marbury T, Dumont E. Pharmacokinetics of Gepotidacin in Renal Impairment. Clin Pharmacol Drug Dev. 2020 Jul;9(5):560-572. doi: 10.1002/cpdd.807. Epub 2020 May 19. PMID 32429000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 2-part study, conducted in participant's with varying degree of renal impairment (RI) which enrolled 32 participants, wherein, 24 participants were enrolled in Part 1 and 8 participants in Part 2. The study was conducted, at 3 centers in United States of America from 29 June 2016 to 20 June 2017.
Pre-assignment Details: A total of 43 participants were screened of which 8 were screen-failures and 32 were enrolled in the study and 3 participants were reserve participants and were no longer required in the study .
Groups:
- Normal, Part 1: The eligible participants, with normal renal function (participants with estimated glomerular filtration rate (eGFR) >= 90 milliliter per minute per 1.73 meter^2 or estimated creatinine clearance (Clcr) >= 90 milliliter per minute), in this arm received a single dose of gepotidacin 750 milligrams, administered as 2-hour intravenous infusion on Day 1.
- Moderate: The eligible participants, with moderate renal function (participants with eGFR in the range of 30 to 59 milliliter per minute per 1.73 meter^2), in this arm received a single dose of gepotidacin at 750 milligrams, administered as 2-hour intravenous infusion on Day 1.
- Severe/ESRD Not on Hemodialysis, Part 1: The eligible participants, with severe renal impairment and participants with ESRD not on hemodialysis renal function (participants with eGFR < 30 milliliter per minute per 1.73 meter^2), in this arm received a single dose of gepotidacin at 750 milligrams, administered as 2-hour intravenous infusion on Day 1.
- ESRD on Hemodialysis, Part 2: The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in this period was separated by a wash-out period of 7-days. These participants, during treatment period 1 on Day 1 and treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour infusion starting approximately 2 hours before the initiation of the last hemodialysis session of the week (Period 1) and gepotidacin 750 milligram, administered as a 2-hour intravenous infusion starting within 2 hours after completion of the last hemodialysis session of the week (treatment period 2).
Period: Part 1 (Up to 44 Days)
Arm/Group | Normal, Part 1 | Moderate | Severe/ESRD Not on Hemodialysis, Part 1 | ESRD on Hemodialysis, Part 2
Started | 8 | 8 | 8 | 0
Completed | 8 | 8 | 8 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 (Up to 50 Days)
Arm/Group | Normal, Part 1 | Moderate | Severe/ESRD Not on Hemodialysis, Part 1 | ESRD on Hemodialysis, Part 2
Started | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal, Part 1: The eligible participants, with normal renal function (participants with estimated glomerular filtration rate (eGFR) >= 90 milliliter per minute per 1.73 meter^2 or estimated Clcr >= 90 milliliter per minute, in this arm received a single dose of gepotidacin 750 milligrams, administered as 2-hour intravenous infusion on Day 1.
- Moderate, Part 1: The eligible participants, with moderate renal function (participants with eGFR in the range of 30 to 59 milliliter per minute per 1.73 meter^2), in this arm received a single dose of gepotidacin at 750 milligrams, administered as 2-hour intravenous infusion on Day 1.
- Total: Total of all reporting groups
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1 | ESRD on Hemodialysis, Part 2 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (10.78) | 72.0 (7.05) | 61.4 (12.49) | 51.8 (7.09) | 61.6 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 1 | 9
  Male | 5 | 7 | 4 | 7 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 2 | 8 | 12
  White: White/Caucasian/European | 7 | 6 | 5 | 0 | 18
  Multiple: African American/African/White | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From Hour 0 to Infinity (AUC[0-inf]) of Gepotidacin for Part 1
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity . Blood samples were collected at the indicated time-points, during the study. The Pharmacokinetic (PK) Parameter Population consisted of all participants in the PK Population, for whom valid and evaluable PK parameters were derived. The PK Population consisted of all participant's, who received at least 1 dose of gepotidacin and had evaluable PK data.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Nanogram*hour per milliliter | 14838 (20.7) | 22367 (17.0) | 28545 (21.4)
Statistical Analysis 1: Comparison: Normal, Part 1 vs Moderate, Part 1; Test type: Other; Ratio of geometric LS means = 1.507, 90% CI 2-sided [0.902 to 2.519] — AUC (0-inf) for participants with normal renal function Vs participants with moderate renal function has been presented
Statistical Analysis 2: Comparison: Normal, Part 1 vs Severe/ESRD Not on Hemodialysis, Part 1; Test type: Other; Ratio of geometric LS means = 1.924, 90% CI 2-sided [1.151 to 3.215] — AUC (0-inf) for participants with normal renal function Vs participants with Severe/ESRD not on hemodialysis

2. Primary Outcome: AUC (0-inf) of Gepotidacin for Part 2
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for gepotidacin. Blood samples were collected at the indicated time-points, during the study.
Time Frame: Pre-dose, 0.25 hours, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose during treatment period 1 and 2 both.
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Groups:
- ESRD on Hemodialysis (Before Hemodialysis), Part 2: The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in each period was separated by a wash-out period of 7-days. These participants, during treatment period 1 on Day 1 and treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour infusion starting approximately 2 hours before the initiation of the last hemodialysis session of the week (treatment period 1).
- ESRD on Hemodialysis (After Hemodialysis), Part 2: The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in each period was separated by a wash-out period of 7-days. These participants, during treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour intravenous infusion starting within 2 hours after completion of the last hemodialysis session of the week (treatment period 2).
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
Nanogram*hour per milliliter | 14838 (20.7) | 35239 (95.0) | 60461 (140.5)
Statistical Analysis 1: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (Before Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 2.375, 90% CI 2-sided [1.421 to 3.969] — AUC (0-inf) for participants with normal renal function Vs ESRD on hemodialysis (before hemodialysis)
Statistical Analysis 2: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (After Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 4.075, 90% CI 2-sided [2.438 to 6.810] — AUC (0-inf) for participants with normal renal function Vs ESRD on hemodialysis (after hemodialysis)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Gepotidacin for Part 1
Description: Cmax, is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples were collected, at the indicated time points for analysis of gepotidacin.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter | 4498 (16.3) | 5306 (16.0) | 7084 (23.3)
Statistical Analysis 1: Comparison: Normal, Part 1 vs Moderate, Part 1; Test type: Other; Ratio of geometric LS means = 1.179, 90% CI 2-sided [0.467 to 2.977] — Cmax for participants with normal renal function Vs participants with moderate renal function has been presented
Statistical Analysis 2: Comparison: Normal, Part 1 vs Severe/ESRD Not on Hemodialysis, Part 1; Test type: Other; Ratio of geometric LS means = 1.575, 90% CI 2-sided [0.624 to 3.975] — Cmax for participants with normal renal function Vs .participants with Severe/ESRD not on hemodialysis

4. Primary Outcome: Cmax of Gepotidacin for Part 2
Description: as for outcome 3
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose on during treatment period 1 and 2 both.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter | 4498 (16.3) | 10123 (216.3) | 26839 (797.1)
Statistical Analysis 1: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (Before Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 2.250, 90% CI 2-sided [0.891 to 5.681] — Cmax for participants with normal renal function Vs ESRD on hemodialysis (before hemodialysis)
Statistical Analysis 2: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (After Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 5.966, 90% CI 2-sided [2.363 to 15.062] — Cmax for participants with normal renal function Vs ESRD on hemodialysis (after hemodialysis)

5. Primary Outcome: Total Amount Excreted in Urine (Ae Total), Part 1
Description: Urine samples from the participants were collected during the study. Ae total assessed the, total unchanged drug (total amount of drug excreted in urine), which was calculated, by adding all the fractions of drug gepotidacin collected, at the indicated time points. No formal statistical analysis of group comparison was planned for urine PK parameters.
Time Frame: Pre-dose (0.0), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose during the single treatment period
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram.
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
milligram. | 280.49 (15.2) | 165.86 (39.4) | 59.40 (68.3)

6. Primary Outcome: Ae Total of Gepotidacin for Part 2
Description: Urine samples, from the participants were collected during the study. Ae total assessed the, total unchanged drug (total amount of drug excreted in urine), which was calculated, by adding all the fractions of drug gepotidacin collected, at the indicated time points. Urine samples were collected at pre-dose (0.0), 0 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose during the single treatment period. Only those participant's available at the specified time points were analyzed. No formal statistical analysis of group comparison was planned for urine PK parameters.
Time Frame: Pre-dose (0.0), 0 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose during both treatment period 1 and 2
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 3 | 3
milligram | 280.49 (15.2) | 7.87 (96.4) | 10.87 (64.7)

7. Primary Outcome: Percentage of the Given Dose Excreted in Urine (fe%) of Gepotidacin for Part 1
Description: The fe% measured the percentage of the given dose of drug gepotidacin, excreted in urine. It was calculated as: Ae total divided by the dose administered multiplied by 100.
Time Frame: At pre-dose (0.0), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose during the single treatment period
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of gepotidacin
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Percentage of gepotidacin | 37.40 (15.2) | 22.11 (39.4) | 7.92 (68.3)

8. Primary Outcome: fe% of Gepotidacin for Part 2
Description: The fe% measured the percentage of the given dose of drug gepotidacin, excreted in urine. It was calculated as: Ae total divided by the dose administered multiplied by 100. No formal statistical analysis of group comparison was planned for urine PK parameters. Only those participants available at the specified time points were analyzed.
Time Frame: At pre-dose (0.0), 0 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose in each of the two treatment periods
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of gepotidacin
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 3 | 3
Percentage of gepotidacin | 37.40 (15.2) | 1.05 (96.4) | 1.45 (64.7)

9. Primary Outcome: Renal Clearance (CLr) of Gepotidacin for Part 1
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time via renal clearance pathways, expressed as volume (Liter) per unit of time (hour). The renal clearance was calculated by Ae total divided by AUC from hour 0 to the last measurable plasma concentration AUC (0-t). Urine samples were collected at pre-dose (0.0), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose during the single treatment period. No formal statistical analysis of group comparison was planned for urine PK parameters.
Time Frame: as for outcome 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Liter per hour | 19.24 (18.8) | 7.58 (44.3) | 2.13 (84.3)

10. Primary Outcome: CLr of Gepotidacin for Part 2
Description: Renal clearance is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time via renal clearance pathways, expressed as volume (Liter) per unit of time (hour). Urine samples were collected at pre-dose (0.0), 0 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours post-dose in each of the two treatment periods. Only those participant's available at the specified time points were analyzed. No formal statistical analysis of group comparison was planned for urine PK parameters.
Time Frame: as for outcome 8
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 3 | 3
Liter per hour | 19.24 (18.8) | 0.29 (101.7) | 0.10 (277.5)

11. Primary Outcome: AUC (t0-t1) of Gepotidacin for Part 2
Description: Partial area under the curve estimated from predialyzer samples collected from start of dialysis (t0) to end of dialysis (t1). Only applicable to Part 2 ESRD on hemodialysis (before hemodialysis) arm..
Time Frame: Dialysate fluid were to be collected on Day 1 after dosing (Period 1 only) at pre-dose from 0 to 4 hours
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 0 | 8 | 0
Nanogram*hour per milliliter |  | 1062 (36.3) |

12. Primary Outcome: Dialysis Clearance (CLD) of Gepotidacin for Part 2
Description: CLD measured the dialysis clearance of gepotidacin over the specified duration in the study and indicates how quickly gepotidacin is cleared out from blood or plasma. Only applicable to Part 2 ESRD on hemodialysis (before hemodialysis) arm.
Time Frame: Pre-dose, 0-1 hours, 1-2 hours, 2-3 hours and 3-4 hours post-dose on Day 1 in Period 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2
Number analyzed (Participants) | 8
Liter per hour | 6.63 (15.8)

13. Primary Outcome: Fraction (%) of the Dose Removed by Hemodialysis From 0 to 4 Hours After the Start of Hemodialysis (Frem%[0-4]) of Gepotidacin for Part 2
Description: Dialysate samples were collected at specified time points in the study. Frem is defined as the fraction (dose in percentage) removed by the process of hemodialysis from 0 to 4 hours after the start of hemodialysis (or to the end of dialysis if less than 4 hours)
Time Frame: Pre-dose, 0-1 hours, 1-2 hours, 2-3 hours and 3-4 hours post-dose on Day 1 in Period 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of gepotidacin removed
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2
Number analyzed (Participants) | 8
Percentage of gepotidacin removed | 5.89 (26.2)

14. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Readings for Part 1
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and corrected Q to T interval (QTc). The data for abnormal ECG recordings not clinically significant (NCS) and clinically significant (CS), have been reported at specific timepoints during the study. No formal analysis of group comparison was planned for dialysate PK parameters
Time Frame: Up to 16 Days
Population: The Safety Population consisted of all participants who received at least 1 dose of study drug and had at least 1 post dose safety assessment.
Measure: Number; unit: Participants
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Baseline, Abnormal, NCS | 3 | 6 | 7
  Baseline, Abnormal, CS | 0 | 0 | 0
  Day 1 - 1.5 hour, Abnormal, NCS | 5 | 6 | 6
  Day 1- 1.5 hour, Abnormal, CS | 0 | 0 | 0
  Day 1- 2 hour, Abnormal, NCS | 3 | 6 | 6
  Day 1- 2 hour, Abnormal, CS | 0 | 0 | 0
  Day 1 - 4 hour, Abnormal, NCS | 2 | 6 | 7
  Day 1- 4 hour, Abnormal CS | 0 | 0 | 0
  Day 1 - 8 hour, Abnormal NCS | 2 | 6 | 6
  Day 1 - 8 hour, Abnormal, CS | 0 | 0 | 0
  Day 1 - 12 hour, Abnormal NCS | 2 | 6 | 7
  Day 1 - 12 hour, Abnormal, CS | 0 | 0 | 0
  Day 2 - 24 hour, Abnormal NCS | 3 | 7 | 5
  Day 2 - 24 hour, Abnormal, CS | 0 | 0 | 0
  Day 2 - 36 hour, Abnormal NCS | 2 | 6 | 6
  Day 2 - 36 hour, Abnormal, CS | 0 | 0 | 0
  Day 3 - 48 hour, Abnormal NCS | 2 | 6 | 5
  Day3 - 48 hour, Abnormal, CS | 0 | 0 | 0
  Follow-up, Abnormal NCS | 3 | 5 | 5
  Follow-up, Abnormal CS | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Abnormal 12-lead ECG Readings for Part 2
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and corrected Q to T interval (QTc). The data for abnormal ECG recordings not clinically significant (NCS) and clinically significant (CS), have been reported at specific time points during the study. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). NA indicates data was not available
Time Frame: Up to 23 Days
Population: Participants
Measure: Number; unit: Participants
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8
Participants
  Day 1- Baseline, Abnormal CS (n=8,8) | 0 | 0
  Day 1 - Baseline, Abnormal NCS (n=8,8) | 6 | 7
  Day 1- 2 hour, Abnormal, NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1- 2 hour, Abnormal, NCS (n=8,0) | 6 |
  Day 1- 2 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1- 2 hour, Abnormal, CS (n=8,0) | 0 |
  Day 1 - 4 hour, Abnormal, NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1 - 4 hour, Abnormal, NCS (n=8,0) | 7 |
  Day 1- 4 hour, Abnormal CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1- 4 hour, Abnormal CS (n=8,0) | 0 |
  Day 1 - 8 hour, Abnormal NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1 - 8 hour, Abnormal NCS (n=8,0) | 7 |
  Day 1 - 8 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1 - 8 hour, Abnormal, CS (n=8,0) | 0 |
  Day 1 - 12 hour, Abnormal NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1 - 12 hour, Abnormal NCS (n=8,0) | 6 |
  Day 1 - 12 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 1 - 12 hour, Abnormal, CS (n=8,0) | 0 |
  Day 2 - 24 hour, Abnormal NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 2 - 24 hour, Abnormal NCS (n=8,0) | 7 |
  Day 2 - 24 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 2 - 24 hour, Abnormal, CS (n=8,0) | 0 |
  Day 2 - 36 hour, Abnormal NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 2 - 36 hour, Abnormal NCS (n=8,0) | 8 |
  Day 2 - 36 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 2 - 36 hour, Abnormal, CS (n=8,0) | 0 |
  Day 3 - 48 hour, Abnormal NCS (n=8,0): number analyzed (Participants) | 8 | 0
  Day 3 - 48 hour, Abnormal NCS (n=8,0) | 7 |
  Day3 - 48 hour, Abnormal, CS (n=8,0): number analyzed (Participants) | 8 | 0
  Day3 - 48 hour, Abnormal, CS (n=8,0) | 0 |
  Day 8- 2 hour, Abnormal, NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8- 2 hour, Abnormal, NCS (n=0,8) |  | 8
  Day 8- 2 hour, Abnormal, CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8- 2 hour, Abnormal, CS (n=0,8) |  | 0
  Day 8 - 4 hour, Abnormal, NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8 - 4 hour, Abnormal, NCS (n=0,8) |  | 8
  Day 8- 4 hour, Abnormal CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8- 4 hour, Abnormal CS (n=0,8) |  | 0
  Day 8 - 8 hour, Abnormal NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8 - 8 hour, Abnormal NCS (n=0,8) |  | 7
  Day 8 - 8 hour, Abnormal, CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8 - 8 hour, Abnormal, CS (n=0,8) |  | 0
  Day 8 - 12 hour, Abnormal NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8 - 12 hour, Abnormal NCS (n=0,8) |  | 8
  Day 8 - 12 hour, Abnormal, CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 8 - 12 hour, Abnormal, CS (n=0,8) |  | 0
  Day 9- 24 hour, Abnormal, NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 9- 24 hour, Abnormal, NCS (n=0,8) |  | 6
  Day 9- 24 hour, Abnormal, CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 9- 24 hour, Abnormal, CS (n=0,8) |  | 0
  Day 9 - 36 hour, Abnormal, NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 9 - 36 hour, Abnormal, NCS (n=0,8) |  | 8
  Day 9- 36 hour, Abnormal CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 9- 36 hour, Abnormal CS (n=0,8) |  | 0
  Day 10 - 48 hour, Abnormal NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 10 - 48 hour, Abnormal NCS (n=0,8) |  | 7
  Day 10 - 48 hour, Abnormal, CS (n=0,8): number analyzed (Participants) | 0 | 8
  Day 10 - 48 hour, Abnormal, CS (n=0,8) |  | 0
  Follow-up, Abnormal NCS (n=0,8): number analyzed (Participants) | 0 | 8
  Follow-up, Abnormal NCS (n=0,8) |  | 6
  Follow-up, Abnormal CS (n=0,8): number analyzed (Participants) | 0 | 8
  Follow-up, Abnormal CS (n=0,8) |  | 0

16. Secondary Outcome: Change From Baseline in Vitals- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure, Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes of rest. The data for change from Baseline values for systolic blood pressure (SBP) and diastolic blood pressure (DBP) was reported. Baseline was defined as the latest pre-dose assessment. Change from Baseline, was defined as post Baseline values minus the values at Baseline.
Time Frame: Baseline and up to 16 Days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter of mercury
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Milliliter of mercury
  SBP, Day 1- 1.5 hour, | 3.1 (2.36) | 6.8 (11.94) | -3.3 (13.77)
  SBP, Day 1- 2 hour, | 6.9 (12.54) | 8.3 (13.39) | -4.4 (12.73)
  SBP, Day 1 - 4 hour | -0.9 (12.15) | 3.4 (5.42) | 1.0 (13.03)
  SBP, Day 1 - 8 hour, | 1.3 (12.69) | 5.9 (7.30) | 6.0 (12.75)
  SBP, Day 1 - 12 hour, | -3.4 (12.29) | 14.1 (12.89) | 4.6 (6.30)
  SBP, Day 2 - 24 hour, | -1.1 (13.28) | 5.3 (6.65) | -4.1 (11.46)
  SBP, Day 2 - 36 hour | 0.5 (3.74) | 14.4 (13.02) | -0.4 (9.12)
  SBP, Day 3 - 48 hour | -1.0 (10.72) | 7.8 (9.10) | -6.0 (18.18)
  SBP, Follow-up | 0.8 (3.28) | 8.3 (13.06) | -4.8 (18.16)
  DBP, Day 1- 1.5 hour | 0.1 (3.91) | -1.3 (3.92) | -3.5 (7.19)
  DBP, Day 1- 2 hour, | 5.8 (7.15) | 1.3 (3.99) | 0.4 (4.07)
  DBP, Day 1 - 4 hour | 3.0 (5.50) | -2.4 (8.14) | 1.5 (4.99)
  DBP, Day 1 - 8 hour | 4.9 (6.06) | -4.3 (10.55) | -2.4 (6.95)
  DBP, Day 1 - 12 hour | 2.9 (6.36) | -0.5 (9.61) | -3.6 (4.66)
  DBP, Day 2 - 24 hour | 2.3 (5.50) | 1.0 (5.55) | -2.3 (4.17)
  DBP, Day 2 - 36 hour | 3.1 (8.22) | -0.8 (13.07) | -3.5 (3.96)
  DBP, Day 3 - 48 hour | 5.0 (7.69) | 0.6 (6.48) | -5.3 (5.87)
  DBP, Follow-up | 2.6 (5.48) | 0.5 (11.60) | -1.8 (6.58)

17. Secondary Outcome: Change From Baseline in Vitals- SBP and DBP, Part 2
Description: Vital signs were measured in semi-supine position after 5 minutes of rest. The data for change from Baseline values for systolic blood pressure (SBP) and diastolic blood pressure (DBP) was reported. Change from Baseline, was defined as post Baseline values minus the values at Baseline. Baseline was defined as the latest pre-dose assessment. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 23 Days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter of mercury
Groups:
- ESRD on Hemodialysis: The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in this period was separated by a wash-out period of 7-days. These participants, during treatment period 1 on Day 1 and treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour infusion starting approximately 2 hours before the initiation of the last hemodialysis session of the week (Period 1) and gepotidacin 750 milligram, administered as a 2-hour intravenous infusion starting within 2 hours after completion of the last hemodialysis session of the week (treatment period 2).
Arm/Group | ESRD on Hemodialysis
Number analyzed (Participants) | 8
Milliliter of mercury
  SBP, Day 1- 2 hour, (n=8) | -0.5 (14.91)
  SBP, Day 1 - 4 hour (n=8) | 8.6 (16.66)
  SBP, Day 1 - 8 hour, (n=8) | -0.6 (23.93)
  SBP, Day 1 - 12 hour, (n=8) | -4.8 (17.68)
  SBP, Day 2 - 24 hour, (n=8) | 1.4 (9.69)
  SBP, Day 2 - 36 hour (n=8) | 3.9 (10.33)
  SBP, Day 3 - 48 hour, (n=8) | 6.5 (5.53)
  SBP, Day 8-2 hour (n=8) | -2.0 (8.16)
  SBP, Day 8-4 hour (n=8) | -4.4 (7.46)
  SBP, Day 8-8 hour (n=8) | -14.8 (14.50)
  SBP, Day 8-12 hour (n=6): number analyzed (Participants) | 6
  SBP, Day 8-12 hour (n=6) | -8.3 (7.92)
  SBP, Day 9-24 hour (n=8) | 5.9 (23.94)
  SBP, Day 9-36 hour (n=8) | 2.3 (20.11)
  SBP, Day 10-48 hour (n=8) | 12.6 (19.72)
  SBP, Follow-up, (n=8) | 0.5 (11.86)
  DBP, Day 1- 2 hour, (n=8) | 4.3 (11.31)
  DBP, Day 1 - 4 hour, (n=8) | 3.6 (9.83)
  DBP, Day 1 - 8 hour, (n=8) | -1.5 (11.70)
  DBP, Day 1 - 12 hour (n=8) | -2.3 (9.54)
  DBP, Day 2 - 24 hour (n=8) | 4.6 (9.68)
  DBP, Day 2 - 36 hour,(n=8) | 3.3 (6.11)
  DBP, Day 3 - 48 hour (n=7): number analyzed (Participants) | 7
  DBP, Day 3 - 48 hour (n=7) | 3.0 (10.10)
  DBP, Day 8-2 hour, (n=8) | -2.1 (10.49)
  DBP, Day 8-4 hour , (n=8) | -2.5 (9.41)
  DBP, Day 8- 8 hour,(n=8) | -6.9 (8.48)
  DBP, Day 8-12 hour, (n=8) | -9.5 (10.03)
  DBP, Day 9-24 hour, (n=8) | 6.4 (9.41)
  DBP, Day 9-36 hour (n=8) | 2.6 (13.41)
  DBP, Day 10-48 hour (n=8) | 5.9 (11.74)
  DBP, Follow-up (n=8) | 2.3 (6.34)

18. Secondary Outcome: Change From Baseline in Vitals- Pulse Rate, Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes of rest. The data for change from Baseline values for pulse rate was reported. Change from Baseline, was defined as post Baseline values minus the values at Baseline. Baseline was defined as the latest pre-dose assessment
Time Frame: Baseline and up to 16 Days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Beats per minute
  Pulse rate, Day 1- 1.5 hour | 0.1 (9.28) | 1.6 (4.21) | 3.5 (4.41)
  Pulse rate, Day 1- 2 hour | 1.8 (7.13) | 4.1 (3.23) | 4.1 (5.03)
  Pulse rate, Day 1 - 4 hour | 0.1 (6.49) | 0.4 (8.14) | 2.0 (5.63)
  Pulse rate, Day 1 - 8 hour | -1.0 (13.40) | 1.8 (7.50) | 0.8 (4.46)
  Pulse rate, Day 1 - 12 hour | -0.1 (12.31) | 3.4 (4.78) | 3.4 (1.92)
  Pulse rate, Day 2 - 24 hour | 1.0 (13.06) | -0.8 (7.85) | -2.3 (5.55)
  Pulse rate, Day 2 - 36 hour | 1.6 (9.56) | -0.5 (5.37) | 0.6 (5.24)
  Pulse rate, Day 3 - 48 hour | -1.4 (10.76) | -0.1 (7.88) | -1.8 (7.34)
  Pulse rate, Follow-up | -0.6 (10.34) | 0.6 (8.45) | 0.0 (7.43)

19. Secondary Outcome: Change From Baseline in Vitals- Pulse Rate, Part 2
Description: Vital signs were measured in semi-supine position after 5 minutes of rest. The data for change from Baseline values for pulse rate was reported. Change from Baseline, was defined as post Baseline values minus the values at Baseline. Baseline was defined as the latest pre-dose assessment. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Up to 23 Days
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | ESRD on Hemodialysis
Number analyzed (Participants) | 8
beats per minute
  Pulse rate, Day 1- 2 hour, (n=8) | 0.4 (8.78)
  Pulse rate, Day 1 - 4 hour, (n=8) | 3.4 (9.09)
  Pulse rate, Day 1 - 8 hour, (n=8) | 4.4 (9.46)
  Pulse rate, Day 1 - 12 hour, (n=7): number analyzed (Participants) | 7
  Pulse rate, Day 1 - 12 hour, (n=7) | 4.4 (10.21)
  Pulse rate, Day 2 - 24 hour, (n=8) | 2.5 (7.11)
  Pulse rate, Day 2 - 36 hour, (n=8) | 6.1 (9.96)
  Pulse rate, Day 3 - 48 hour, (n=7): number analyzed (Participants) | 7
  Pulse rate, Day 3 - 48 hour, (n=7) | 3.6 (5.88)
  Pulse rate, Day, 8-2 hour (n=8) | 4.8 (10.38)
  Pulse rate, Day 8-4 hour (n=7): number analyzed (Participants) | 7
  Pulse rate, Day 8-4 hour (n=7) | 2.1 (5.08)
  Pulse rate, Day 8-8 hour ,(n=8) | 3.4 (7.69)
  Pulse rate, Day 8-12 hour (n=8) | 4.7 (10.05)
  Pulse rate, Day 9-24 hour (n=8) | 4.0 (11.51)
  Pulse rate, Day9-36 hour (n=8) | 8.9 (16.19)
  Pulse rate, Day 10-48 hour (n=8) | 3.6 (11.04)
  Pulse rate, Follow-up (n=8) | 3.8 (10.22)

20. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs) for Part 1
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: Up to 16 Days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Any SAE | 0 | 0 | 0
  Any AE | 0 | 3 | 4

21. Secondary Outcome: Number of Participants With Any AEs and Any SAEs for Part 2
Description: as for outcome 20
Time Frame: Up to 23 Days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8
Participants
  Any SAE | 0 | 0
  Any AE | 4 | 3

22. Secondary Outcome: Number of Participants With Clinical Laboratory Test Results for Grade 3 or Higher for Part 1
Description: The adverse events reported by the participants were classified as Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe) and Grade 4 as life-threatening. The data for clinical laboratory findings with values of Grade 3 or higher, have been reported.
Time Frame: Up to 17 Days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Serum or plasma creatinine, Grade 3 or higher | 0 | 0 | 5
  Serum glucose, Grade 3 or higher | 0 | 0 | 1

23. Secondary Outcome: Number of Participants With Clinical Laboratory Test Results for Grade 3 or Higher for Part 2
Description: as for outcome 22
Time Frame: Up to 24 Days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8
Participants
  Serum or plasma creatinine, Grade 3 or higher | 8 | 0
  Serum glucose, Grade 3 or higher | 2 | 0

24. Secondary Outcome: Number of Participants With Abnormal Physical Examination Results for Part 1
Description: Physical exam were to be performed by a qualified individual. A complete physical examination included, at a minimum, an assessment of the cardiovascular, respiratory, GI, and neurological systems. Height and weight were also measured and recorded. A brief physical examination included, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). This data was not collected.
Time Frame: Up to 16 Days
Population: Safety Population. This data was not collected.
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Abnormal Physical Examination Results for Part 2
Description: as for outcome 24
Time Frame: Up to 23 Days
Population: Safety Population: This data was not collected.
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: AUC (0-t) of Gepotidacin for Part 1
Description: Blood samples were collected at specified time-points for PK analysis. The data for Area under the concentration-time curve from time 0 (predose) to time of last quantifiable concentration for gepotidacin were reported.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Nanogram*hour per milliliter | 14582 (20.8) | 21883 (17.1) | 27886 (21.4)
Statistical Analysis 1: Comparison: Normal, Part 1 vs Severe/ESRD Not on Hemodialysis, Part 1; Test type: Other; Ratio of geometric LS means = 1.501, 90% CI 2-sided [0.894 to 2.520] — Normal Vs Moderate
Statistical Analysis 2: Comparison: Normal, Part 1 vs Severe/ESRD Not on Hemodialysis, Part 1; Test type: Other; Ratio of geometric LS means = 1.912, 90% CI 2-sided [1.139 to 3.212] — Normal Vs Severe/ESRD not on hemodialysis

27. Secondary Outcome: AUC (0-t) of Gepotidacin for Part 2
Description: Serial blood samples were collected at specified time-points for PK analysis. The data for Area under the concentration-time curve from time 0 (predose) to time of last quantifiable concentration for gepotidacin were reported.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose during treatment period 1 and 2 both.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
Nanogram*hour per milliliter | 14582 (20.8) | 34633 (95.8) | 59311 (143.3)
Statistical Analysis 1: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (Before Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 2.375, 90% CI 2-sided [1.414 to 3.989] — Normal Vs ESRD on hemodialysis (before hemodialysis)
Statistical Analysis 2: Comparison: Normal, Part 1 vs ESRD on Hemodialysis (After Hemodialysis), Part 2; Test type: Other; Ratio of geometric LS means = 4.068, 90% CI 2-sided [2.422 to 6.831] — Normal Vs ESRD on hemodialysis (after hemodialysis)

28. Secondary Outcome: Systemic Clearance (CL) of Gepotidacin for Part 1
Description: Serial blood samples were collected at specified time-points for PK analysis. Systemic CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma AUC(0-inf).
Time Frame: At pre-dose and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose during the single treatment period.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Liter per hour | 50.55 (20.7) | 33.53 (17.0) | 26.27 (21.4)

29. Secondary Outcome: CL of Gepotidacin for Part 2
Description: as for outcome 28
Time Frame: At pre-dose and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose in each of the two treatment periods
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
Liter per hour | 50.55 (20.7) | 21.28 (95.0) | 12.40 (140.5)

30. Secondary Outcome: Terminal Elimination Rate Constant (lambda_z) of Gepotidacin for Part 1
Description: Serial blood samples were collected at specified time-points for PK analysis. It is the ratio of clearance to volume of distribution and is expressed in units of 1/hour.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Per hour | 0.06027 (11.9) | 0.06369 (16.1) | 0.06266 (13.4)

31. Secondary Outcome: Lambda_z of Gepotidacin for Part 2
Description: as for outcome 30
Time Frame: as for outcome 4
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Per hour | 0.06027 (11.9) | 0.07338 (8.4) | 0.06428 (16.4)

32. Secondary Outcome: Terminal Phase Half-life (t1/2) of Gepotidacin for Part 1
Description: Serial blood samples were collected at specified time-points for PK analysis. t1/2 is defined as the time required by the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
hours | 11.663 [9.549 to 13.065] | 11.421 [7.402 to 12.259] | 11.246 [8.901 to 14.046]

33. Secondary Outcome: t1/2 of Gepotidacin for Part 2
Description: as for outcome 32
Time Frame: as for outcome 27
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
hours | 11.663 [9.549 to 13.065] | 9.455 [8.441 to 10.915] | 11.121 [8.275 to 12.896]

34. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Gepotidacin for Part1
Description: Serial blood samples were collected at specified time-points for PK analysis. Tmax was defined as the time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: Pharmacokinetic Parameter Population
Measure: Mean (Full Range); unit: hours
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
hours | 2.000 [1.00 to 2.00] | 2.000 [1.50 to 2.00] | 2.000 [0.25 to 2.50]

35. Secondary Outcome: Tmax of Gepotidacin for Part 2
Description: as for outcome 34
Time Frame: as for outcome 27
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
hours | 2.000 [1.00 to 2.00] | 2.000 [0.50 to 2.02] | 1.575 [0.25 to 2.00]

36. Secondary Outcome: Volume of Distribution at Steady State of Parent Drug (Vss) of Gepotidacin for Part 1
Description: Serial blood samples were collected at specified time-points for PK analysis. Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Liter | 255 (21.7) | 223 (14.8) | 181 (23.5)

37. Secondary Outcome: Vss of Gepotidacin for Part 2
Description: as for outcome 36
Time Frame: as for outcome 27
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
Liter | 255 (21.7) | 114 (335.6) | 49 (938.8)

38. Secondary Outcome: Volume of Distribution of the Terminal Phase (Vz) of Gepotidacin for Part 1
Description: Serial blood samples were collected at specified time-points for PK analysis. Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vz is the apparent volume of distribution at terminal phase. Volume of distribution of the terminal phase was calculated as total administered dose of gepotidacin divided by AUC (0-inf) multiplied by the rate constant.
Time Frame: Pre-dose, 0.25 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8 | 8
Liter | 839 (25.3) | 527 (29.1) | 419 (27.0)

39. Secondary Outcome: Vz of Gepotidacin for Part 2
Description: as for outcome 38
Time Frame: as for outcome 27
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 8 | 8
Liter | 839 (25.3) | 290 (90.8) | 193 (161.3)

40. Secondary Outcome: Cumulative Amount of Drug Excreted in Urine From Time t1 to t2 (Ae[t1-t2]) of Gepotidacin for Part 1, for Normal
Description: Ae (t1-t2), measure the amount of drug excreted in urine in a time intervals for predose, 0 to 6, 6 to 12, 12 to 24, or 24 to 36, and 36 to 48 hours after dosing for participant's with renal impairment; and predose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours for participant's with normal renal function.
Time Frame: At Pre-dose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Normal, Part 1
Number analyzed (Participants) | 8
milligram
  Ae(0-2) | 135.53 (21.0)
  Ae (2-4) | 59.95 (56.7)
  Ae (4-6) | 19.90 (18.4)
  Ae (6-8) | 19.47 (70.5)
  Ae (8-12) | 9.11 (86.9)
  Ae(12-24) | 12.30 (55.3)
  Ae(24-36) | 5.38 (52.1)
  Ae(36-48) | 3.00 (42.8)

41. Secondary Outcome: Cumulative Amount of Drug Excreted in Urine From Time t1 to t2 (Ae[t1-t2]) of Gepotidacin for Part 1, for Moderate and Severe
Description: Ae (t1-t2), measure the amount of drug excreted in urine in a time intervals for predose, 0 to 6, 6 to 12, 12 to 24, or 24 to 36, and 36 to 48 hours after dosing for participant's with renal impairment. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: at pre-dose (0.0), 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 36, and 36 to 48 hours post-dose during the single treatment period
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1
Number analyzed (Participants) | 8 | 8
milligram
  Ae (0-6) (n=8, 8) | 119.79 (50.0) | 39.54 (94.9)
  Ae (6-12) (n=8, 8) | 21.67 (30.7) | 8.26 (44.8)
  Ae (12-24) (n=8, 8) | 12.81 (40.8) | 4.42 (160.0)
  Ae(24-36 (n=8, 8) | 5.25 (25.4) | 2.89 (29.8)
  Ae(36-48) (n=8,7): number analyzed (Participants) | 8 | 7
  Ae(36-48) (n=8,7) | 2.66 (50.3) | 1.17 (71.0)

42. Secondary Outcome: Ae(t1-t2) of Gepotidacin for Part 2
Description: Ae (t1-t2), measure the amount of drug excreted in urine in a time intervals for predose, 0 to 6, 6 to 12, 12 to 24, or 24 to 36, and 36 to 48 hours after dosing for participant's with renal impairment; and predose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours for participant's with normal renal function. NA indicates data is not available due to insufficient participants.Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 6
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Normal, Part 1 | ESRD on Hemodialysis (Before Hemodialysis), Part 2 | ESRD on Hemodialysis (After Hemodialysis), Part 2
Number analyzed (Participants) | 8 | 3 | 3
milligram
  Ae (0-8)(n=0,3,3): number analyzed (Participants) | 0 | 3 | 3
  Ae (0-8)(n=0,3,3) |  | 5.56 (123.4) | 8.12 (73.8)
  Ae (8-12) (n=8,3,3) | 9.11 (86.9) | 0.72 (32.1) | 1.16 (31.5)
  Ae (12-24) (n=8,3, 3) | 12.30 (55.3) | 0.81 (147.5) | 1.31 (52.5)
  Ae (24-36) (n=8,2,1): number analyzed (Participants) | 8 | 2 | 1
  Ae (24-36) (n=8,2,1) | 5.38 (52.1) | 0.45 (154.4) | 0.75 (NA) — NA indicates data is not available due to insufficient participants".
  Ae (36-48) (n=8,2,0): number analyzed (Participants) | 8 | 2 | 0
  Ae (36-48) (n=8,2,0) | 3.00 (42.8) | 0.14 (133.2) |

43. Secondary Outcome: Total Amount of Unchanged Amount of Drug Removed by Hemodialysis (Arem) From Time 0 to 1 Hour After the Start of Hemodialysis (Arem[0-1]), Arem (1-2), Arem (2-3), Arem (3-4) for Part 2
Description: Arem is defined as the total amount of drug removed using the hemodialysis method at different timepoints namely Arem (0-1), measured the amount of drug removed by hemodialysis from time 0 to 1 hour after the start of hemodialysis; Arem (1-2), measured the amount of drug removed by hemodialysis from time 1 to 2 hours after the start of hemodialysis; Arem(2-3) ), measured the amount of drug removed by hemodialysis from time 2 to 3 hour, Arem (3-4), measured the amount of drug removed by hemodialysis from hemodialysis from time 3 to 4 hours after the start of hemodialysis (or to the end of dialysis if <4 hours). Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0-1 hours, 1-2 hours, 2-3 hours and 3-4 hours post-dose on Day 1 in Period 1Dialysate fluid were collected at 1, 2, 3, and 4 hours post-dose in Period 1 only
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | ESRD on Hemodialysis (Before Hemodialysis), Part 2
Number analyzed (Participants) | 8
milligram
  Arem (0-1), (n=8) | 18.22 (27.7)
  Arem (1-2), (n=8) | 12.42 (34.8)
  Arem (2-3), (n=8) | 8.93 (32.5)
  Arem (3-4), (n=6): number analyzed (Participants) | 6
  Arem (3-4), (n=6) | 5.35 (36.6)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of study treatment upto 94 days
Description: AEs and SAEs were collected in Safety Population.
Groups:
- ESRD on Hemodialysis (Before Hemodialysis): The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in each period was separated by a wash-out period of 7-days. These participants, during treatment period 1 on Day 1 and treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour infusion starting approximately 2 hours before the initiation of the last hemodialysis session of the week (treatment period 1).
- ESRD on Hemodialysis (After Hemodialysis): The participants in this arm, in the part 2 of the study participated in 2 treatment periods. The dosing in each period was separated by a wash-out period of 7-days. These participants, during treatment period 2 on Day 8, received a single dose of study drug gepotidacin 750 milligram, administered as a 2-hour intravenous infusion starting within 2 hours after completion of the last hemodialysis session of the week (treatment period 2).
Arm/Group | Normal, Part 1 | Moderate, Part 1 | Severe/ESRD Not on Hemodialysis, Part 1 | ESRD on Hemodialysis (Before Hemodialysis) | ESRD on Hemodialysis (After Hemodialysis)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 4/8 | 4/8 | 4/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal, Part 1 (N=8) | Moderate, Part 1 (N=8) | Severe/ESRD Not on Hemodialysis, Part 1 (N=8) | ESRD on Hemodialysis (Before Hemodialysis) (N=8) | ESRD on Hemodialysis (After Hemodialysis) (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Infusion site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02729038/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT02729038/SAP_001.pdf